CLINICAL TRIAL: NCT05528601
Title: Observational Study on the Influence of an App-based Self-management Program on the Quality of Life of Women With Endometriosis
Brief Title: Influence of an App on Quality of Life of Women With Endometriosis
Acronym: pre ELEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Dr. med. Sebastian Daniel Schäfer, PI, University Hospital Muenster
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pre ELEA
Record Dates: First submitted 2022-08-18; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Endometriosis; Quality of Life
Keywords: endometriosis; quality of life; smartphone application
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: two arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- users (Experimental): app users
  Interventions: Behavioral: use of Endo App®
- non-users (No Intervention): app non-users

INTERVENTIONS:
Behavioral: use of Endo App® — use of Endo App® smartphone application containing endometriosis relevant exercises and educational material
  Arms: users

SUMMARY:
Comparison of quality of life before and after 14 days of use of Endo App® in endometriosis patients compared to non-users

DETAILED DESCRIPTION:
Introduction: Endometriosis can significantly impair the quality of life of those affected. Multimodal self-help measures are recommended but often difficult to access. Smartphone apps have been shown to improve quality of life for other conditions with chronic pain. The aim of this study was to examine whether there is evidence of beneficial effects of the Endo-App and whether a multicenter randomized controlled trial should be planned to substantiate these effects.

Methods: In a sample of N=106 women affected by endometriosis the present study determined the influence of the use of a smartphone app (Endo-App ®) on their quality of life. Among others, the validated questionnaire Endometriosis Health Profile from Oxford University was used for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* suffering from endometriosis
* 18 years or older
* willing and capable of using a smartphone

Exclusion Criteria:

* minor under 18 years
* endometriosis excluded
* not capable of using a smartphone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — applicable for participants with female body
Enrollment: 106 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
quality of life of endometriosis patients | 14 days
  quality of life measured bei Endometriosis Health Profile 30

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Münster Germany, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rohloff N, Rothenhofer M, Gotz T, Schafer SD. Observational pilot study on the influence of an app-based self-management program on the quality of life of women with endometriosis. Arch Gynecol Obstet. 2024 Aug;310(2):1157-1170. doi: 10.1007/s00404-024-07468-4. Epub 2024 Jun 13. PMID 38869629